CLINICAL TRIAL: NCT06061393
Title: Comparison Between Outcomes of Pregnant Women Treated With Ferinject vs. Venofer for Iron Deficiency Anemia (Hb<9)
Brief Title: Comparison Between Outcomes of Pregnant Women Treated With Ferinject vs. Venofer for Iron Deficiency Anemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, Principal Investigator., Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-23-NHR
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Anemia, Iron Deficiency; Pregnancy Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferric Oxide, Saccharated; Injections; ferric carboxymaltose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- venofer (Active Comparator): Women with iron def. anemia aith hemoglobin level <9 gr/dl who will be traeted with venofer
  Interventions: Drug: Venofer 200 MG Per 10 ML Injection
- Ferinject (Active Comparator): Women with iron def. anemia aith hemoglobin level <9 gr/dl who will be traeted with ferinject
  Interventions: Drug: Ferinject

INTERVENTIONS:
Drug: Venofer 200 MG Per 10 ML Injection — treat anemia with venofer up to 5 doses
  Arms: venofer
Drug: Ferinject — ferinject 500 mg, once a week for 2 weeks
  Arms: Ferinject

SUMMARY:
The purpose of this study is to compare maternal outcomes such as increased hemoglobin need for blood transfusion and hemoglobin level before and post partum in women with hemoglobin <9 gr/dl , treated with venofer and women treated with ferinject.

ELIGIBILITY:
Inclusion Criteria:

pregnancy>24 weeks of gestation anemia with Hb<8 anemia with Hb<9 if symptomatic anemia of previous postpartum hemorrhage

Exclusion Criteria:

* Allergy to one of the study's drugs
* IV iron treatment in the last month
* chronic anemia- thalassemia, renal failure Twins pregnancy
* non iron deficiency anemia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 200 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
ratio of women with Hb level >11 at delivery | at delivery
  Hb level
postpartum Hb level | during 48 hours after delivery
  gr/dl